CLINICAL TRIAL: NCT00286936
Title: Incidence of Delirium in Hip Fracture Patients Randomized to Regular Hypnotics vs Placebo
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow inclusion resulting in premature termination due to logistics
Sponsor: Hvidovre University Hospital (Other)
Collaborators: IMK Fonden (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HHSG-RCT-05
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2006-09

CONDITIONS: Hip Fracture; Delirium
Keywords: Hip fracture; delirium; sleep disturbance; hypnotic
MeSH Terms: conditions — Hip Fractures; Delirium; Parasomnias | interventions — Zolpidem

INTERVENTIONS:
Drug: Zolpidem

SUMMARY:
To examine the influence of regular hypnotic therapy on the incidence of delirium after hip fracture surgery

DETAILED DESCRIPTION:
Delirium is prevalent after hip fracture surgery. Delirium has been linked to postoperative sleep disturbances. Zolpidem is a non-benzodiazepine hypnotic that preserves REM sleep. The present study investigates the incidence of delirium in hip fracture patients randomized to Zolpidem treatment 5 mg vs placebo in the perioperative phase.

ELIGIBILITY:
Inclusion Criteria:

* Primary hip fracture, no substance abuse, no regular opioid, corticosteroid or benzodiazepine therapy, hepatic insufficiency, myastenia gravis, allergies to drug components

Exclusion Criteria:

* Severe respiratory insufficiency

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2004-02; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of postoperative delirium

SECONDARY OUTCOMES:
Sleep quality
mobilization
loss of functional ability
length of stay
sedation
nocturnal nursing events

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai B Foss, MD, Study Director — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark